CLINICAL TRIAL: NCT02302859
Title: Mobile Smoking Cessation Treatment for Underserved Smokers: A Pilot and Feasibility Study
Brief Title: Mobile Media-Rich Interactive Guideline System (MMRIGS) Pilot Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: At the request of the PI
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2014-0509; NCI-2014-02572 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2014-11-21; First posted 2014-11-27 (Estimated); Results first posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Tobacco Use Cessation
Keywords: Cancer Prevention; Tobacco Use Cessation; HIV-positive; Nicotine patch; NRT; Questionnaire; Survey; Smartphone; Counseling; Saliva test; Saliva cotinine test; Nicotine replacement therapy; Smoking abstinence; Aids
MeSH Terms: conditions — Tobacco Use Cessation; HIV Seropositivity; Acquired Immunodeficiency Syndrome | interventions — Tobacco Use Cessation Devices; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Treatment (ST) (Experimental): Participants supplied with a 8-week supply of nicotine patches, a smart phone and brief advice to quit smoking. Participants also receive proactive phone counseling (8 sessions) over the 8-week period for support in quitting smoking. The call will last about 15 minutes.
  Participants receive weekly assessments to complete for the 8-week treatment period via smartphone.
  Participants receive weekly assessments to complete for the 8-week treatment period via smartphone, and again at 3 months after intervention.
  Participants complete saliva cotinine test 3 months after intervention.
  Interventions: Drug: Nicotine Patch; Behavioral: Questionnaires; Other: Pamphlet; Behavioral: Phone Counseling Sessions; Other: Saliva Test; Device: Smart phone
- Automated Treatment (AT) (Experimental): Participants supplied with a 8-week supply of nicotine patches and a smart phone. Participants also receive brief advice to quit smoking (tailored video clips) and an 8-week automated intervention (interactive text messages and graphical messages) for support in quitting smoking via smartphone.
  Participants receive weekly assessments to complete for the 8-week treatment period via smartphone, and again at 3 months.
  Participants complete saliva cotinine test 3 months after intervention.
  Interventions: Drug: Nicotine Patch; Behavioral: Questionnaires; Behavioral: Phone Counseling Sessions; Other: Saliva Test; Device: Smart phone

INTERVENTIONS:
Drug: Nicotine Patch — Participants receive an 8 week supply of Nicotine patches.
  Other Names: NRT
Behavioral: Questionnaires — Questionnaire completion at baseline on laptop, then weekly for 8 weeks on smartphone, then 3 months after smartphone intervention.
  Other Names: Surveys
Other: Pamphlet — Pamphlet given to participant describing health and financial reasons to quit smoking.
  Arms: Standard Treatment (ST)
Behavioral: Phone Counseling Sessions — Standard Treatment (ST) Group: Participants receive 8 phone counseling sessions (one session per week) for support in quitting smoking. The calls should last about 15 minutes.
  Automated Treatment (AT) Group: Participants receive brief video clips with advice on how to quit smoking over smartphone, as well as interactive text and picture messages once a week for 8 weeks. The video clips will be about 5 minutes long.
  Participants also have access to additional counseling content on the smart phone, which can be used at any time.
Other: Saliva Test — Participants complete saliva cotinine test 3 months after intervention.
Device: Smart phone — Standard Treatment (ST) Group: Participants receive proactive phone counseling (8 sessions) over the 8-week period for support in quitting smoking. The call will last about 15 minutes.
  Automated Treatment (AT) Group: Participants receive brief advice to quit smoking (tailored video clips) and an 8-week automated intervention (interactive text messages and graphical messages) for support in quitting smoking via smartphone.

SUMMARY:
The goal of this research study is to learn about 2 different interactive methods that are designed to help people with HIV/AIDS stop smoking.

DETAILED DESCRIPTION:
Baseline Questionnaire:

If you agree to take part in this study, you will complete a questionnaire on a laptop about your feelings, mood, health, thoughts about smoking, thoughts about quitting smoking, smoking history, and some demographic information such as age, education level, and income level. This should take about 15-20 minutes to complete.

Study Groups:

After completing the questionnaire, you will be randomly assigned (as in the flip of a coin) to 1 of 2 study groups. You will have an equal chance of being placed in either group.

Both groups will receive smart phones and an 8-week supply of nicotine patches with instructions on how to use them. Each group will receive different methods of advice for quitting smoking.

If you are assigned to Group 1, the following study procedures will be performed:

* You will receive brief advice on how to quit smoking once at the time of enrollment. The advice will be given from a pamphlet that has information such as health problems related to smoking, how many Americans are affected each year, financial problems related to smoking, nicotine replacement therapy options, preparation for quitting smoking, and encouragement to quit.
* On the smart phone, you will have 5 phone counseling sessions for support in quitting smoking throughout the 8-week intervention treatment. The calls should last about 15 minutes.

If you are assigned to Group 2, the following study procedures will be performed:

* On the smart phone, you will receive brief video clips with advice on how to quit smoking, as well as interactive text and picture messages once a week for 8 weeks. The video clips will be about 5 minutes long.
* You will also have access to additional counseling content on the smart phone, which you can use at any time.

Weekly Smart Phone Questionnaires:

Both groups will complete questionnaires on the smart phone every week for 8 weeks. Each questionnaire will have questions about your current smoking status, your motivation level to stop smoking, and things that may have a negative effect on your quitting. The questionnaire should take about 15 minutes to complete.

Follow-up Saliva Test and Questionnaire:

About 3 months after your first smart phone intervention, both groups will complete a saliva test and take a photograph of the test results. The saliva test results will be used to check your smoking activity. Supplies and instructions will be given to you when you are enrolled on the study and the instructions will be available on the smart phone. You will also complete a questionnaire similar to the baseline questionnaire.

Length of Study:

You will be on study for about 3 months.

This is an investigational study. Up to 50 participants will take part in this study. All will be enrolled at the Harris Health System (Thomas Street Health Center).

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Smoked at least 100 cigarettes in lifetime
3. English speaking
4. HIV-positive patient at Thomas Street Health Center
5. Currently smoking 5 or more cigarettes per day
6. Willing to make a quit attempt within 1 week of enrollment

Exclusion Criteria:

1. Positive history of a medical condition that precludes use of the nicotine patch
2. Current use of nicotine replacement therapy (NRT)
3. Current use of other smoking cessation medications (e.g., Chantix or Zyban)
4. Pregnant or nursing
5. Enrolled in another smoking cessation study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diana S. Hoover, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- Thomas Street Health Center -Harris Health System, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period Opened January 2015 and Closed March 2016. Recruitment was accomplished in clinic setting of a large comprehensive HIV-care center.
Groups:
- Standard Treatment (ST): Participants receive 15-minute proactive weekly phone counseling sessions via smartphone along with supply of nicotine patches for 8-week period to support quitting smoking.
- Automated Treatment (AT): Participants receive brief weekly advice (tailored 5 minute video clips) and 8-week automated intervention (interactive text messages and graphical messages via smartphone) along with supply of nicotine patches for 8-week period to support quitting smoking.
Period: Overall Study
Arm/Group | Standard Treatment (ST) | Automated Treatment (AT)
Started | 2 | 6
Completed | 1 | 4
Not Completed | 1 | 2
Not completed — Lost Phone | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Treatment (ST) | Automated Treatment (AT) | Total
Number analyzed (Participants) | 2 | 6 | 8
Age, Continuous [Median (Full Range); unit: years] | 46 [44 to 48] | 54 [44 to 57] | 51 [44 to 57]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 0 | 4 | 4
Region of Enrollment [Number; unit: participants]
  United States | 2 | 6 | 8

OUTCOME MEASURES:

1. Primary Outcome: Smoking Abstinence: 3-month Assessment Via Smart Phone
Description: Smoking abstinence defined as number of participants with biochemically 7-day abstinence confirmed with weekly smart-phone assessments. Saliva cotinine levels, assessed with NicAlert test strips, used to biochemically verify abstinence. Participants will complete the NicAlert saliva cotinine test (supplies given at enrollment) and take a photograph of the test strip results. In primary abstinence analysis for difference in cessation rate between interventions, participants who do not complete follow-up assessments considered to be smokers.
Time Frame: 3 months
Population: Data were not collected due to early termination of the protocol
Arm/Group | Standard Treatment (ST) | Automated Treatment (AT)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data collected over 3 month treatment period.
Arm/Group | Standard Treatment (ST) | Automated Treatment (AT)
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/6
Other Adverse Events (participants affected / at risk) | 0/2 | 0/6

LIMITATIONS AND CAVEATS:
Early termination leading to small number of subjects registered, study halted without analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes